CLINICAL TRIAL: NCT06471192
Title: Predictors of Thrombus Burden in STEMI Patients and Their Impact on Outcome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaaeldin Abdelrahman, Dr, Assiut University
Other Study IDs: predictors of thrombus burden
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: PPCI — PPCI for patients of STEMI to assess thrombus burden

SUMMARY:
ST-segment elevation myocardial infarction (STEMI) is the most acute manifestation of coronary artery disease and is associated with great morbidity and mortality.(1). High thrombus burden (HTB) during ST-segment elevation myocardial infarction (STEMI) could translate into worse clinical outcomes.(2). HTB has been defined as the occurrence of thrombo- sis during myocardial infarction, as determined by a thrombus score ≥ 3 in the infarct-related artery (IRA) or as a "cut-off" occlusion pattern and/or large reference vessel diameter (≥ 3.5 mm) in an occluded IRA.(3) Many variables were used to predict the presence of high thrombus burden in STEMI patients undergoing primary PCI. higher C-reactive protein, and low serum albumin, higher C - reactive protein to albumin ratio (4) which can be used as a surrogate marker of pro-inflammation and is closely related to pro-thrombotic state. Furthermore higher neutrophil-lymphocyte ratio is closely associated with HTB and short-term mortality in STEMI patients (5). MAPH score, which is a new score that combines blood viscosity biomarkers such as mean platelet volume (MPV), total protein and hematocrit, can be used to predict thrombus burden in ST-segment elevation myocardial infarction (STEMI) patients.(6). In addition, TyG index, a valid surrogate marker of insulin resistance, is an independent predictor of LTB in STEMI patients who underwent primary PCI and can be used as an indicator of increased intracoronary thrombus burden. (7). Furthermore, Initial troponin level may be associated with larger thrombus burden within a coronary artery. This finding may influence coronary flow and needs to be taken into consideration during primary coronary intervention.(8). The atherogenic index, a logarithmically transformed ratio of molar concentrations of triglycerides to HDL-cholesterol, can be used as a reliable marker for increased coronary thrombus burden, which is associated with adverse cardiovascular outcomes(9).whole blood viscosity has also been showing that WBV at both shear rates is a significant predictor of HTB in NSTEMI patients(10).

In our research, we aim to study the effect of these different parameters on thrombus burden and their impact on patients outcome at 6 months

DETAILED DESCRIPTION:
ST-segment elevation myocardial infarction (STEMI) is the most acute manifestation of coronary artery disease and is associated with great morbidity and mortality.(1). High thrombus burden (HTB) during ST-segment elevation myocardial infarction (STEMI) could translate into worse clinical outcomes.(2). HTB has been defined as the occurrence of thrombo- sis during myocardial infarction, as determined by a thrombus score ≥ 3 in the infarct-related artery (IRA) or as a "cut-off" occlusion pattern and/or large reference vessel diameter (≥ 3.5 mm) in an occluded IRA.(3) Many variables were used to predict the presence of high thrombus burden in STEMI patients undergoing primary PCI. higher C-reactive protein, and low serum albumin, higher C - reactive protein to albumin ratio (4) which can be used as a surrogate marker of pro-inflammation and is closely related to pro-thrombotic state. Furthermore higher neutrophil-lymphocyte ratio is closely associated with HTB and short-term mortality in STEMI patients (5). MAPH score, which is a new score that combines blood viscosity biomarkers such as mean platelet volume (MPV), total protein and hematocrit, can be used to predict thrombus burden in ST-segment elevation myocardial infarction (STEMI) patients.(6). In addition, TyG index, a valid surrogate marker of insulin resistance, is an independent predictor of LTB in STEMI patients who underwent primary PCI and can be used as an indicator of increased intracoronary thrombus burden. (7). Furthermore, Initial troponin level may be associated with larger thrombus burden within a coronary artery. This finding may influence coronary flow and needs to be taken into consideration during primary coronary intervention.(8). The atherogenic index, a logarithmically transformed ratio of molar concentrations of triglycerides to HDL-cholesterol, can be used as a reliable marker for increased coronary thrombus burden, which is associated with adverse cardiovascular outcomes(9).whole blood viscosity has also been showing that WBV at both shear rates is a significant predictor of HTB in NSTEMI patients(10).

In our research, we aim to study the effect of these different parameters on thrombus burden and their impact on patients outcome at 6 months

Study tools(in detail, e.g., lab methods, instruments, steps, chemicals, …):

A-History taking:

Patients' data will be collected, included age, gender and comorbidities.

B- physical examination including:

* Waist -to-hip ratio
* Body mass index (BMI)
* Waist circumference
* Systolic, diastolic and mean blood pressure C- Laboratory investigations
* Complete blood picture (CBC)
* S. Urea, S. Creatinine (Cr), uric acid (UA), S. Sodium, S. Potassium
* S.troponin
* Cpk,Cpk mb
* lipid profile
* Blood glucose levels at time of admission ,during hospitalization and at discharge
* CRP
* HbA1c
* S.total protein, S. ALB D- 12 lead ECG E-Score and ratio calculations A- MAPH score The predictive cut-off values of MPV, total protein, age and hematocrit for high thrombus grade were determined using the Youden index. The values higher from the cut-off were considered as a score of 1 and MAPH score was calculated as the sum score of 0 or 1 by the cut-off in each ratio.(6).

B- CRP/albumin ratio SA and CRP levels are obtained from the results of blood samples taken immediately during admission to the emergency department. CAR values were obtained by dividing the CRP level by the SA level.(4).

C- Tri-glycerides glucose index TyG index is calculated as ln [fasting triglycerides (mg/dL) × fasting plasma glucose (mg/dL).(7).

D- Neutrophil-to-lymphocyte ratio Complete blood count is obtained from taken immediately during admission to the emergency department.NLR values were obtained by dividing the neutrophil count by lymphocyte count.(5).

E- Atherogenic index The atherogenic index is calculated by using the following formula: log10 (TG/HDL-C)7 and classified as follows: 0.3 to 0.1 indicated a low risk, 0.1 to 0.24 indicated a medium risk, and more than 0.24 indicated a high risk of CVD. (9).

F- Whole blood viscosity WBV at a high shear rate (HSR) (208 sec-1) and a low shear rate (LSR) (0.5 sec-1) were determined using HTC (percent) and total protein (g/l) levels; WBV at HSR (208 sec-1) = (0.12 × HTC) + (0.17 × [total protein-2.07]) and WBV at LSR (0.5 sec-1) = (1.89 × HTC) + (3.76 × [total protein-78.42]) (10)

E-Angiographic analysis for determination of thrombus burden:

The angiographic data will be revised by two experienced interventional cardiologists. Intracoronary thrombus at baseline are angiographically identified and scored according to Thrombolysis in Myocardial Infarction (TIMI) thrombus grade (11). grade 0 (G0) no angiographic characteristics of thrombus are present; grade 1 (G1) possible thrombus is present, with angiographic characteristics as reduced contrast density, haziness, irregular lesion contour, or a smooth convex meniscus, suggestive but not diagnostic of thrombus; grade 2 (G2) there is definite thrombus with greatest dimensions 1/2 or less of the vessel diameter; grade 3 (G3) there is definite thrombus with greatest linear dimension greater than 1/2 but less than 2 vessel diameters; grade 4 (G4) there is definite thrombus with the largest dimension at least 2 vessel diameters; grade 5 (G5) there is total occlusion.

F. Type of stent G. Echocardiography: for assessment of left side function systolic and diastolic function, right side systolic function & valvular affection.

All echocardiographic measurements will be performed according to the recommendations of the American Society of Echocardiography using a high -resolution Phillips machine.

H. In hospital MACE

A total of 0 to 3 points on the HEART score is considered low risk, with a risk of 0.6% to 1.7% for major adverse cardiac events (MACE) in the four to six weeks after presentation. A score of 4 to 6 is intermediate risk (16.6% risk of MACE), and 7 to 10 points is high risk (50.1% risk of MACE). (12)

Clinical follow-up:

Information about the survival status of all patients through hospital records and contact with patients and their relatives.

Information on hospitalization and cardiovascular events will be obtained through health questionnaires. If necessary, referring cardiologists and general practitioners were contacted for additional data. In case of re-hospitalization medical records or discharge letters from other hospitals will be collected. Clinical follow-up was performed at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted with STEMI undergoing PPCI will be recruited in the study and the period of data collection will be continued for 12 months. Total number that will be recruited will be at least 200 cases.

Exclusion Criteria:

* known chronic inflammatory disease, neoplasms or severe hepatic disease; end-stage renal disorder (estimated glomerular filtration rate < 30 ml/min/1.73 m2); undergoing renal replacement therapy; no intracoronary lesions shown via angiography; history of cardiac valve surgery; using oral anticoagulants;

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted with STEMI undergoing PPCI will be recruited in the study and the period of data collection will be continued for 12 months. Total number that will be recruited will be at least 200 cases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect different factors on thrombus burden in patients with STEMI. | 1 year
  To evaluate the effect different factors on thrombus burden in patients with STEMI.

SECONDARY OUTCOMES:
Impact of these factors on patients outcomes at 6 months. | 18 months
  Impact of these factors on patients outcomes at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Soheir Kasem, Professor, Study Director — Soher.Kasem@yahoo.com

IPD SHARING:
Plan to Share IPD: Undecided